CLINICAL TRIAL: NCT05672147
Title: Phase I Study of Cellular Immunotherapy Using T Cells Lentivirally Transduced to Express a Cd33-Specific Chimeric Antigen Receptor for Patients With Cd33+ Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: CD33-CAR T Cell Therapy for the Treatment of Recurrent or Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21665; NCI-2022-10310 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21665 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia; Recurrent Adult Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (anti-CD33 CAR T-cells) (Experimental): Patients undergo lymphodepletion therapy 3-5 days prior to CAR T cell infusion and receive anti-CD33 CAR T-cells IV on day 0. Patients with persistent CD33+ AML who are > 28 days past the initial CAR T infusion, have additional product available and did not experience a dose-limiting toxicity, may optionally receive anti-CD33 CAR T-cells IV.
  Interventions: Biological: Anti-CD33 CAR T-cells; Procedure: Lymphodepletion Therapy

INTERVENTIONS:
Biological: Anti-CD33 CAR T-cells — Given IV
  Other Names: Anti-CD33 CAR T Cells; Anti-CD33 CAR-T Cells; CD33-CAR T Cells
Procedure: Lymphodepletion Therapy — Undergo lymphodepletion
  Other Names: Lymphodepleting Therapy; Lymphodepletion

SUMMARY:
This phase I trial tests the safety, side effects, and the best dose of anti-CD33 chimeric antigen receptor (CAR) T-Cell therapy in treating patients with acute myeloid leukemia that has come back (recurrent) or does not respond to treatment (refractory). CAR T-cell therapy is a type of treatment in which a patient or donor's T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T cells are taken from a patient's or donor's blood. Then the gene for a special receptor that binds to a certain protein on the patient's cancer cells is added to the T cells in the laboratory. The special receptor is called a chimeric antigen receptor. Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Examine the anti-tumor activity and safety of administering patient-specific donor-derived (allogeneic) CD33-CAR T cells following lymphodepletion in research participants with CD33+ recurrent/refractory (r/r) acute myeloid leukemia (AML).

SECONDARY OBJECTIVE:

I. Assess activity in the form of CAR T cell expansion and persistence, to assess impact on hematopoiesis, 6-month progression free survival (PFS 6mo) rate, duration of response, and 1-year overall survival (OS) rate.

EXPLORATORY OBJECTIVES:

I. Change from baseline in numbers of CD33+ blood cells, CD33 expression on leukemia cells and hematopoietic cells.

II. For subjects who receive cetuximab for CAR T cell ablation, assess the activity of infusional cetuximab to eliminate transferred CD33R(CD8h)BBzeta/EGFRt+ T cells.

OUTLINE: This is a dose-escalation study.

Patients undergo lymphodepletion therapy 3-5 days prior to CAR T cell infusion and receive anti-CD33 CAR T-cells intravenously (IV) on day 0. Patients with persistent CD33+ AML who are > 28 days past the initial CAR T infusion, have additional product available and did not experience a dose-limiting toxicity, may optionally receive anti-CD33 CAR T-cells IV.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
  * For research participants who do not speak English, a short form consent may be used with a City of Hope (COH) certified interpreter/translator to proceed with screening, while the request for a translated full consent is processed
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with Study principal investigator (PI) approval
* Age: >= 18 years
* Karnofsky Performance Scale (KPS) >= 70
* Life expectancy >= 16 weeks at the time of enrollment
* Prior allogeneic transplant allowed if > 6 months prior to study enrollment
* Participant must have a confirmed diagnosis of active CD33+ AML de novo, or secondary OR participants who are at a high risk for disease recurrence

  * Relapsed AML is defined as patients that had a first complete response (CR) before developing recurrent disease (increased bone marrow blasts)
  * Refractory AML is defined as patients that have not achieved a first CR after induction chemotherapy. For patients with AML evolving from myelodysplastic syndrome, they should have completed at least one cycle of induction chemotherapy
* Research participants must have bone marrow and/or peripheral blood samples available for confirmation of diagnosis of AML

  * CD33 positivity must be confirmed by either flow cytometry or immunohistochemistry within 90 days of study entry. Cytogenetics, flow cytometry, and molecular studies (such as FLT-3 status) will be obtained as per standard practice
  * Research participants who are at a high risk of disease recurrence, they must have historical bone marrow and/or peripheral blood samples available for confirmation of diagnosis of AML
* No known contraindications to lymphodepleting agents, steroids, tocilizumab and/or cetuximab, or the investigational agent
* Total serum bilirubin =< 2.0 mg/dL
* Participants with Gilbert syndrome may be included if their total bilirubin is =< 3.0
* Aspartate aminotransferase (AST) =< 3 x the upper limit of normal (ULN)
* Alanine aminotransferase (ALT) =< 3 x ULN
* Estimated creatinine clearance of >= 60 mL/min per the Cockcroft-Gault formula, and the participant is not on hemodialysis
* Left ventricular ejection fraction >= 50% within 8 weeks before enrollment
* Oxygen (O2) saturation > 92% not requiring oxygen supplementation
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test
* If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* Research participants must have a potential donor or stem cell source identified for allogeneic transplantation, either related (7/8 or 8/8 allele matched or haploidentical)
* DONOR: The identified donor must be the original donor whose stem cells were used for the research participant's allogeneic hematopoietic stem cell transplantation (alloSCT)
* DONOR: The donor must be HIV negative
* DONOR: KPS >= 70
* DONOR: Documented body weight

Exclusion Criteria:

* Prior allogeneic transplant if < 6 months prior to enrollment
* Concurrent use of systemic steroids or chronic use of immunosuppressant medications should be stopped 28-days prior to enrollment. Recent or current use of inhaled or topical steroids in standard doses is not exclusionary. Physiologic replacement of steroids (prednisone =< 7.5 mg/day, or equivalent doses of other corticosteroids) is allowed
* Participants with active autoimmune disease, including graft versus host disease (GvHD), requiring systemic immune suppressive should be stopped 28-days prior to enrollment
* Participants may not be receiving any other investigational agents and are not dependent on concurrent biological therapy, chemotherapy, or radiation therapy

  * With exception to Hydrea which must be stopped prior to initiation of lymphodepletion
* Research participants on active systemic antifungal treatment within 8 weeks of enrollment are not eligible. However, participants on antifungal prophylaxis are eligible

  * Not applicable at the time of enrollment if the research participant's donor is undergoing leukapheresis
* Subjects with >= Grade 2 myelofibrosis on bone marrow biopsy
* Subjects with clinically significant arrhythmia or arrhythmias not stable on medical management within two weeks of screening if the patient is undergoing leukapheresis. Patients with controlled atrial arrythmia is allowed
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 6 months prior to screening
* Subjects with presence of other active malignancy, however, research participants with history of prior malignancy treated with curative intent and in complete remission are eligible
* Clinically significant uncontrolled illness
* Active infection requiring antibiotics
* Research participants who have tested human immunodeficiency virus (HIV) positive, or have active hepatitis B or C infection based on testing performed within 4 weeks of enrollment
* Active viral hepatitis
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2028-09-03 (Estimated); Study Completion 2028-09-03 (Estimated)

PRIMARY OUTCOMES:
Participants who achieve measurable residual disease (MRD) | Up to 15 years post study treatment
  Defined as complete response (CR) or MRD- complete response with incomplete hematopoietic recovery. Rates and associated 90% Clopper and Pearson binomial confidence limits.
Incidence of dose-limiting toxicities and full toxicity profile | Up to 1 year following the last CAR T cell infusion
  Rates and associated 90% toxicity and adverse events will be assessed using Common Terminology Criteria for Adverse Events version 5.0, and modified Cytokine Release Syndrome grading as applicable. Clopper and Pearson binomial confidence limits.

SECONDARY OUTCOMES:
Expansion and persistence of the CAR T cell product | Up to 15 years post-CAR T cell infusion
  Descriptive statistics and graphical methods will be used to present expansion and persistence.
Percent and counts from peripheral blood cell subsets in hematopoietic stem/progenitor cell compartments | Up to 15 years post-CAR T cell infusion
  Descriptive statistics and graphical methods will be used to present T cell numbers and percentages over time.
Duration of response | From the first achievement of CR after CAR T cell infusion through disease relapse or progression or death, assessed up to 15 years post CAR T cell infusion
  Patients who have not had disease relapse/progression or death at the last follow-up will be censored at the time of last follow-up. Patients who never achieved CR will be excluded from the analysis. Descriptive statistics will be provided for duration of response.
Progression-free survival | From the start of treatment to the date of death, disease relapse, or last follow-up whichever occurs first, assessed up to 15 years post CAR T cell infusion
  Participants are considered a failure for this endpoint if they die (regardless of cause) or experience disease relapse.
Overall survival | from start of protocol therapy to death, or last follow-up, whichever comes first, assessed up to 15 years post CAR T cell infusion
  Participants are considered a failure for this endpoint if they die, regardless of cause.

CONTACTS AND LOCATIONS:
Overall Officials: Karamjeet S Sandhu, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States